CLINICAL TRIAL: NCT06872073
Title: Assessment of Methotreaxate-induced Liver Fibrosis by Transient Elastography and Serological Markers
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, heba ali Mohammed, Residant doctor, Assiut University
Other Study IDs: MTX liver fibrosis TE
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Liver Fibrosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: patients prescribed Methotrexate therapy for Rheumatological disease (such as Systemic Lupus Erythematosus , Rheumatoid arthritis and Ankylosing spondylitis)or Dermatological diseases (such as Psoriasis and Behcets disease).
- Group B: patients with Rheumatological or Dermatological disease who have not received Methotrexate

SUMMARY:
Methotrexate (MTX), a folic acid analogue, inhibits the synthesis of purines and pyrimidines and is widely used in the treatment of chronic inflammatory diseases, particularly Rheumatoid arthritis (RA). It is typically the first-line drug for RA management. However, prolonged MTX use is associated with hepatotoxicity, including liver fibrosis (LF), which necessitates regular monitoring, especially of liver function tests MTX-induced liver injury has been recognized since the early 1970and numerous studies have shown an increased risk of liver fibrosis, which is estimated to occur in approximately 5% of patients, with a potential relationship to the cumulative dose of MTX Despite intensive monitoring strategies and the recommendation for liver biopsies, liver biopsy carry significant risk, including bleeding and sampling variability .

the aim of the study to Estimate the frequency and stage of liver fibrosis in patients with Rheumatological or Dermatological diseases receiving Methotrexate in Assuit University Hospitals in comparison to a control group with the same diseases not receiving Methotrexate.

Evaluate the diagnostic performance of FIB-4 , APRI and FIB-5 scores as non invasive fibrosis markers in comparison to Transient Elastography in these patients.

Identify the predictors of liver fibrosis in these patients. As such, there is increasing interest in non-invasive methods for monitoring liver fibrosis, such as liver stiffness measurement by FibroScan (FS), APRI score , FIB-4 score and FIB-5 score . These methods offer advantages over liver biopsy, including being non-invasive, rapid, reproducible, and able to assess disease progression over time. However, the prevalence of hepatic fibrosis in MTX-treated patients, particularly in Egypt, remains under-researched.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) prescribed Methotrexate therapy for Rheumatological disease (such as Systemic Lupus Erythematosus , Rheumatoid arthritis and Ankylosing spondylitis)or Dermatological diseases (such as Psoriasis and Behcets disease).

Exclusion Criteria:

* Patients with metabolic associated fatty liver disease (MAFLD). Patients with chronic liver diseases (HBV, HCV, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, alcoholic liver disease).

History of chronic heart failure or renal failure.c.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults (18 years and older) prescribed Methotrexate therapy for Rheumatological disease (such as Systemic Lupus Erythematosus , Rheumatoid arthritis and Ankylosing spondylitis)or Dermatological diseases (such as Psoriasis and Behcets disease).
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
prevelance of liver fibrosis | baseline
  Estimate the frequency of liver fibrosis in patients with Rheumatological or Dermatological diseases receiving Methotrexate in Assuit University Hospitals